CLINICAL TRIAL: NCT03104686
Title: Pasta and Bread Prepared With Durum Wheat Semolina: Effect on Post-prandial Glucose and Insulin Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Francesca Scazzina Ph.D., Assistant Professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pane2
Record Dates: First submitted 2017-02-28; First posted 2017-04-07 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Desiccation; Bread; Glucose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Personnel involved in randomization, in the analyses of the samples collected, and who were involved in the data processing were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bread (Active Comparator): Bread (50g available carbohydrate, 109 g) eaten with 500 mL of water
  Interventions: Other: Bread
- Short pasta (dry) (Experimental): Cooked penne (142 g; 71 g uncooked) eaten with 500 mL of water
  Interventions: Other: Short pasta (dry)
- Long pasta (dry) (Experimental): Cooked spaghetti (142 g; 71 g uncooked) eaten with 500 mL of water
  Interventions: Other: Long pasta (dry)
- Glucose (Active Comparator): Glucose monohydrate (55 g) dissolved with 500 mL of water
  Interventions: Other: Glucose

INTERVENTIONS:
Other: Short pasta (dry) — 50g available carbohydrate of penne pasta
  Other Names: Penne
  Arms: Short pasta (dry)
Other: Long pasta (dry) — 50g available carbohydrate of spaghetti pasta
  Other Names: Spaghetti
  Arms: Long pasta (dry)
Other: Bread — 50g available carbohydrate of bread
  Arms: Bread
Other: Glucose — 50g available carbohydrate of glucose monohydrate
  Arms: Glucose

SUMMARY:
Carbohydrate-based products can influence the post-prandial glycemic response differently based on their ability to be digested, absorbed and to affect rises in plasma glucose. Pasta is one of the major carbohydrate-rich foods consumed in Italy. Studies from the literature describe a lower glycemic response after the consumption of pasta compared with other wheat-based products, such as bread. Among the factors affecting post-prandial glycemia after consumption of carbohydrate-based products, the technological process represents a central one. In fact, the different technological processes alter the food matrix which can affect the post-prandial metabolism of glucose and insulin differently. Thus, the present study aims at investigating the effect induced by the principal steps of the process of pasta production on the reduction of post-prandial glycemic and insulinemic responses.

DETAILED DESCRIPTION:
The different glycemic responses after the consumption of carbohydrate-based products are associated with different rates of digestion and absorption of the carbohydrates in the human body. Therefore, food products rich in carbohydrates can be classified based on their ability to be digested, absorbed and to affect post-prandial glycemia. Epidemiological studies suggest that following a diet including carbohydrate-based foods inducing a low and slow glycemic response is associated with reduced risk to develop some non-communicable diseases (such as type 2 diabetes and cardiovascular disease), to control inflammatory status, which is the trigger of several pathologies, and to reduce fasting insulin. Depending on the food composition, a low glycemic response is not always associated with a low plasma insulin concentration. For instance, high protein or lipid concentrations in the food matrix have been demonstrated to induce low post-prandial glycemic responses, but not a reduction in insulin secretion. Avoiding a high insulin post-prandial response after consumption of foods represents a preventive factor against the risk of overweight and hyperlipidemia, type 2 diabetes, and cancer. Therefore, the evaluation of both glycemic and insulinemic post-prandial response curves is necessary in order to demonstrate the true beneficial effect of the consumption of low glycemic index foods. Among several factors which can influence the post-prandial glycemic and insulinemic responses (such as macronutrient composition and the cooking process), the technological aspects through which the foods are produced represent an important one. Several studies reported a low glycemic response after the consumption of pasta compared with bread, and this is due to the technological structures characterizing the two matrices. Pasta is one of the major sources of carbohydrates consumed in Italy. Therefore, the aim of the present study is to investigate the effect of pasta and bread on the plasma response of glucose and insulin, as well as c-peptide in order to clearly discriminate the different biological effect induced by the technological process in the production of pasta, compared to foods beginning with the same ingredients. Moreover, the study aims to create a solid basis for future studies for evaluating the effect of pasta consumption, as the main source of carbohydrates, in a context of a balanced diet, for maintaining health.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female

Exclusion Criteria:

* BMI>30kg/m2
* celiac disease
* metabolic disorders (diabetes, hypertension, dislipidemia, glucidic intolerance)
* chronic drug therapies for any pathologies (including psychiatric diseases)
* intense physical activity
* dietary supplements affecting the metabolism
* anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
incremental area under the curve for blood glucose | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  postprandial response for blood glucose (IAUC)
incremental area under the curve for plasma insulin | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  postprandial response for plasma insulin (IAUC)

SECONDARY OUTCOMES:
post-prandial c-peptide plasma concentration | 2 hours (-10 and 0 -fasting-, 15, 30, 45, 60, 90, 120 minutes)
  postprandial response for plasma c-peptide (IAUC)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Scazzina, PhD, Principal Investigator — Department of Food Science, University of Parma; Furio Brighenti, PhD, Study Director — Department of Food Science, University of Parma
Locations (1):
- Department of Food Science, University of Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blaak EE, Antoine JM, Benton D, Bjorck I, Bozzetto L, Brouns F, Diamant M, Dye L, Hulshof T, Holst JJ, Lamport DJ, Laville M, Lawton CL, Meheust A, Nilson A, Normand S, Rivellese AA, Theis S, Torekov SS, Vinoy S. Impact of postprandial glycaemia on health and prevention of disease. Obes Rev. 2012 Oct;13(10):923-84. doi: 10.1111/j.1467-789X.2012.01011.x. Epub 2012 Jul 11. PMID 22780564
- [Background] Collier GR, Greenberg GR, Wolever TM, Jenkins DJ. The acute effect of fat on insulin secretion. J Clin Endocrinol Metab. 1988 Feb;66(2):323-6. doi: 10.1210/jcem-66-2-323. PMID 3276722
- [Background] Dong JY, Zhang L, Zhang YH, Qin LQ. Dietary glycaemic index and glycaemic load in relation to the risk of type 2 diabetes: a meta-analysis of prospective cohort studies. Br J Nutr. 2011 Dec;106(11):1649-54. doi: 10.1017/S000711451100540X. Epub 2011 Sep 29. PMID 22017823
- [Background] Gannon MC, Nuttall FQ, Neil BJ, Westphal SA. The insulin and glucose responses to meals of glucose plus various proteins in type II diabetic subjects. Metabolism. 1988 Nov;37(11):1081-8. doi: 10.1016/0026-0495(88)90072-8. PMID 3054432
- [Background] Jenkins DJ, Wolever TM, Jenkins AL. Starchy foods and glycemic index. Diabetes Care. 1988 Feb;11(2):149-59. doi: 10.2337/diacare.11.2.149. PMID 3383733
- [Background] Jenkins DJ, Wolever TM, Taylor RH, Barker H, Fielden H, Baldwin JM, Bowling AC, Newman HC, Jenkins AL, Goff DV. Glycemic index of foods: a physiological basis for carbohydrate exchange. Am J Clin Nutr. 1981 Mar;34(3):362-6. doi: 10.1093/ajcn/34.3.362. PMID 6259925
- [Background] Livesey G, Taylor R, Livesey H, Liu S. Is there a dose-response relation of dietary glycemic load to risk of type 2 diabetes? Meta-analysis of prospective cohort studies. Am J Clin Nutr. 2013 Mar;97(3):584-96. doi: 10.3945/ajcn.112.041467. Epub 2013 Jan 30. PMID 23364021
- [Background] Ludwig DS. The glycemic index: physiological mechanisms relating to obesity, diabetes, and cardiovascular disease. JAMA. 2002 May 8;287(18):2414-23. doi: 10.1001/jama.287.18.2414. PMID 11988062
- [Background] Ma XY, Liu JP, Song ZY. Glycemic load, glycemic index and risk of cardiovascular diseases: meta-analyses of prospective studies. Atherosclerosis. 2012 Aug;223(2):491-6. doi: 10.1016/j.atherosclerosis.2012.05.028. Epub 2012 Jun 6. PMID 22727193
- [Background] Onitilo AA, Stankowski RV, Berg RL, Engel JM, Glurich I, Williams GM, Doi SA. Type 2 diabetes mellitus, glycemic control, and cancer risk. Eur J Cancer Prev. 2014 Mar;23(2):134-40. doi: 10.1097/CEJ.0b013e3283656394. PMID 23962874
- [Background] Ostlund RE Jr, Staten M, Kohrt WM, Schultz J, Malley M. The ratio of waist-to-hip circumference, plasma insulin level, and glucose intolerance as independent predictors of the HDL2 cholesterol level in older adults. N Engl J Med. 1990 Jan 25;322(4):229-34. doi: 10.1056/NEJM199001253220404. PMID 2403660
- [Background] Petitot, M., Abecassis, J. & Micard, V. Structuring of pasta components during processing: impact on starch and protein digestibility and allergenicity. Trends Food Sci Tech. 2009;20,521-532
- [Background] Schwingshackl L, Hoffmann G. Long-term effects of low glycemic index/load vs. high glycemic index/load diets on parameters of obesity and obesity-associated risks: a systematic review and meta-analysis. Nutr Metab Cardiovasc Dis. 2013 Aug;23(8):699-706. doi: 10.1016/j.numecd.2013.04.008. Epub 2013 Jun 17. PMID 23786819
- [Background] Sieri S, Krogh V, Berrino F, Evangelista A, Agnoli C, Brighenti F, Pellegrini N, Palli D, Masala G, Sacerdote C, Veglia F, Tumino R, Frasca G, Grioni S, Pala V, Mattiello A, Chiodini P, Panico S. Dietary glycemic load and index and risk of coronary heart disease in a large italian cohort: the EPICOR study. Arch Intern Med. 2010 Apr 12;170(7):640-7. doi: 10.1001/archinternmed.2010.15. PMID 20386010
- [Background] Weyer C, Funahashi T, Tanaka S, Hotta K, Matsuzawa Y, Pratley RE, Tataranni PA. Hypoadiponectinemia in obesity and type 2 diabetes: close association with insulin resistance and hyperinsulinemia. J Clin Endocrinol Metab. 2001 May;86(5):1930-5. doi: 10.1210/jcem.86.5.7463. PMID 11344187
- [Background] Wolever TM, Jenkins DJ, Kalmusky J, Giordano C, Giudici S, Jenkins AL, Thompson LU, Wong GS, Josse RG. Glycemic response to pasta: effect of surface area, degree of cooking, and protein enrichment. Diabetes Care. 1986 Jul-Aug;9(4):401-4. doi: 10.2337/diacare.9.4.401. PMID 3743316
- [Derived] Vanhatalo S, Dall'Asta M, Cossu M, Chiavaroli L, Francinelli V, Pede GD, Dodi R, Narvainen J, Antonini M, Goldoni M, Holopainen-Mantila U, Cas AD, Bonadonna R, Brighenti F, Poutanen K, Scazzina F. Pasta Structure Affects Mastication, Bolus Properties, and Postprandial Glucose and Insulin Metabolism in Healthy Adults. J Nutr. 2022 Apr 1;152(4):994-1005. doi: 10.1093/jn/nxab361. PMID 34669959